CLINICAL TRIAL: NCT06356870
Title: Alveolar Cleft Reconstruction Using BMAC and Allograft vs Iliac Cancellous Bone: A Randomized Clinical Trial.
Brief Title: Alveolar Cleft Reconstruction Using Bone Marrow Aspirate Concentrate and Allograft vs Iliac Cancellous Bone.
Acronym: BMAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Moustafa Ismail Abdelmaksoud, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUE
Record Dates: First submitted 2024-03-30; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Alveolar Cleft Grafting
Keywords: BMAC; alveolar cleft
MeSH Terms: interventions — Transplantation, Homologous

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allograft mixed with BMAC (Experimental): Allograft mixed with BMAC used for alveolar cleft grafting
  Interventions: Procedure: BMAC MIXED WITH ALLOGRAFT
- Anterior iliac crest cancellous bone only (Active Comparator): Anterior iliac crest cancellous bone only used for alveolar cleft grafting
  Interventions: Procedure: Cancellous bone from anterior iliac crest

INTERVENTIONS:
Procedure: BMAC MIXED WITH ALLOGRAFT — Study group
  Arms: Allograft mixed with BMAC
Procedure: Cancellous bone from anterior iliac crest — Control group
  Arms: Anterior iliac crest cancellous bone only

SUMMARY:
radiographic and clinical assessment of alveolar cleft grafting using Allograft mixed with BMAC compared to the standard protocol of anterior iliac crest cancellous bone grafting

DETAILED DESCRIPTION:
In the study group BMAC is collected after processing of bone marrow aspirated from anterior iliac crest using a stab incision and a specialized trocar with no surgical intervention at donor site. The BMAC will be mixed with allow graft and used for alveolar cleft grafting

In the control group the standard protocol for alveolar cleft grafting will be used which is surgical exposure of the anterior iliac crest and harvesting of cancellous bone particles.

ELIGIBILITY:
Inclusion Criteria:

* alveolar cleft patients at the mixed dentition phase

Exclusion Criteria:

* patients with previous alveolar grafting intervention

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
bone density | 6 months
  Assessment of bone density at the grafting site from a CT scan using Hounsfild Unit (HU)

SECONDARY OUTCOMES:
Bone gain | 6 months
  Assessment of bone gain at the grafting site from a CT scan in millimeters
Postoperative donor site morbidity | 1 month
  Assessment of donor site morbidity with a questionnaire (VAS Score)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No